CLINICAL TRIAL: NCT06750354
Title: A Randomized Controlled Study to Evaluate the Effect of Papworth Technique and Aerobic Training on Hemoglobin and Exercise Tolerance in Anemic Asthmatic Pediatrics
Brief Title: Study on Effect of Papworth Technique in Anemic Asthmatic Pediatrics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alshaimaa Alsayed Ali, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005437
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Anaemia; Asthma Exacerbations
Keywords: papworth technique; aerobic training; anaemic asthmatic pediatrics
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Patients will be included:
  1. 40 patients from both genders.
  2. Participants between the age 12 and 18 years
  3. Oriented, medically stable and taking their medical treatment
  4. Mild and moderate asthma
  5. All patients are diagnosed as iron deficiency anemia
  6. Body mass index between 18.5 -24.9
  While excluded if:
  1. Have any serious chest diseases, Patients with heart diseases.
  2. Patients with neurological disease affecting respiratory muscles or any muscular dystrophy
  3. Patients with kidney diseases
  4. Patients with liver diseases
  5. Other types of anaemia Chest deformities
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): will receive papworth technique and aerobic training programme in addition to medical treatment 3 sessions per week for 12 weeks.
  Interventions: Procedure: papworth technique; Procedure: aerobic training
- Control group (Active Comparator): aerobic training programme only in addition to medical treatment3 sessions per week for 12 weeks
  Interventions: Procedure: aerobic training

INTERVENTIONS:
Procedure: papworth technique — For Group A: The Papworth breathing technique consists of a series of diaphragmatic breathing and relaxation exercises, and teaches patients which muscles to use when breathing and how to avoid breathing too or too fast by emphasizing nose breathing. The technique is altered to suit activity; this allows the technique to be integrated by patients into their everyday lives with subsequent improvements in quality of life.
  Arms: Study group
Procedure: aerobic training — Aerobic training exercises are any activities that raise heart rate and make breathing somewhat harder. The activity you are doing must be constant and continuous. Examples of aerobic activities are
  Walking or hiking Jogging or running Biking Swimming Rowing In-line skating Cross-country skiing Exercising on a stair-climber or elliptical machine

SUMMARY:
As asthma is chronic condition which interferes with quality of life and exercise tolerance, so it is important to find out cost-effective alternative for the management of asthma due to increased prevalence and rising health care cost as well . Therefore, to provide comprehensive asthma treatment, it is necessary to rule out and address the factor affecting quality of life and exercise tolerance. Asthmatics require stepwise approach which contains assessment treatment planning and review of response. Along with this modification of risk factors, controller therapy is adjusted accordingly. But this is inadequate for asthma management as pharmacological management has some side effects. So, in addition to medical care, Papworth method provides good adjuvant to control asthma symptoms. Asthma subjects require comprehensive approach to deal with these hyperinflation and hyperventilation which are common manifestations of asthma

DETAILED DESCRIPTION:
PURPOSE: This study will be conducted to detect the effect of papworth technique and aerobic training on haemoglobin and exercise tolerance in anaemic asthmatic pediatrics

BACKGROUND: One of the chronic inflammatory diseases is asthma, which manifests symptoms like breathlessness, coughing, wheezing, and chest tightness also, commonly at night or in the early morning. Papworth method is easy and safe intervention for asthma control as it is also an adjuvant to medical care. Papworth method reduces these asthma symptoms, improves dysfunctional breathing arising from hypocapnia, and will help in improving quality of life and exercise tolerance.

HYPOTHESESThere is no significant effect of papworth technique and aerobic training on haemoglobin in anaemic asthmatic pediatrics there is no significant effect of papworth technique and aerobic training on exercise tolerance in anaemic asthmatic pediatricsas regards to:

1. Haemoglobin level
2. Asthma-related Quality of life questionnaire (AQLQ)
3. Six-minute walk test.
4. Oxygen saturation
5. Respiratory rate RESEARCH QUESTION: Is there is an effect of papworth technique and aerobic training on haemoglobin and exercise tolerance in anaemic asthmatic pediatrics?

Patients will be assessed before, after the treatment program. The assessment procedures include the following items:

1. Haemoglobin level
2. asthma-related Quality of life questionnaire (AQLQ)
3. Six-minute walk test.
4. Oxygen saturation
5. Respiratory rate

Treatment procedure:

Group (A): will receive papworth technique and aerobic training programme in addition to medical treatment 3 sessions per week for 12 weeks.

Group (B): will receive aerobic training programme only in addition to medical treatment3 sessions per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included:

1. 40 patients from both genders.
2. Participants between the age 12 and 18 years
3. Oriented, medically stable and taking their medical treatment
4. Mild and moderate asthma
5. All patients are diagnosed as iron deficiency anemia
6. Body mass index between 18.5 -24.9

Exclusion Criteria:

1. Have any serious chest diseases, Patients with heart diseases. 2. Patients with neurological disease affecting respiratory muscles or any muscular dystrophy 3. Patients with kidney diseases 4. Patients with liver diseases 5. Other types of anaemia Chest deformities

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin level | AFTER 12 WEEKS
  Oxygen saturation measures how much hemoglobin is bound to oxygen compared to how much hemoglobin remains unbound.
  a normal pulse oximeter reading for your oxygen saturation level is between 95% and 100%
Asthma-related Quality of life questionnaire (AQLQ) | AFTER 12 WEEKS
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item questionnaire used to assess the physical, occupational, emotional, and social qualities of adults aged 17 to 70 years with asthma.
  The AQLQ has 4 domains: symptoms (12 items), activity limitation (6 generic and 5 patient-specific items), emotional function (5 items), and environmental stimuli (4 items). The AQLQ was developed for patients exhibiting mild to moderate asthma. The AQLQ items are each scored on a 7-point Likert scale, with 1 representing maximal impairment and 7 representing no impairment.
Six-minute walk test. | AFTER 12 WEEKS
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility.
Oxygen saturation | AFTER 12 WEEKS
  by using a normal pulse oximeter reading for your oxygen saturation level is between 95% and 100%. If you have a lung disease such as COPD or pneumonia, your normal oxygen saturation level may be lower.
Respiratory rate | AFTER 12 WEEKS
  The normal respiratory rate for healthy adults is between 12-20 breaths per minute. At this breathing rate, the carbon dioxide exits the lungs at the same rate that the body produces it. Breathing rates of below 12 or above 20 can mean a disruption in the breathing processes.

IPD SHARING:
Plan to Share IPD: No